CLINICAL TRIAL: NCT02162992
Title: Repolarization Disorders and Heart Conduction Disorders in Patients With Systemic Lupus Erythematous
Brief Title: Systemic Lupus Erythematous and Heart Conduction Disorders
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Roger Villuendas Sabaté, Coordinator of the Electrophysiology and Cardiac Pacing Unit, Germans Trias i Pujol Hospital
Other Study IDs: ICOR-2014-01
Record Dates: First submitted 2014-04-24; First posted 2014-06-13 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Lupus Erythematosus, Systemic; Atrioventricular Block; Sudden Death
Keywords: Antibodies, Antinuclear; SS-A antigen; Lupus Erythematosus, Systemic; Atrioventricular Block; Sudden death
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atrioventricular Block; Death, Sudden

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SLE and Anti-Ro antibodies Group: Patients with SLE visited in the rheumatology outpatient's area. No intervention (only observational)
  Interventions: Other: No intervention
- SLE without Anti-Ro antibodies Group: Patients with SLE visited in the rheumatology outpatient's area. No intervention (only observational)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational

SUMMARY:
Connective tissue diseases have been related to heart conduction disorders. The anti-Ro/SSA antibodies are thought to have a pathogenic role, and they most prevalent in systemic lupus erythematous (SLE). The aim of this study is to evaluate the relationship between SLE, arrhythmias and its serologic profile.

DETAILED DESCRIPTION:
We designed a cross-sectional study for an observational analysis. The target population will be the group of SLE patients visited the service of Rheumatology hospitals in Catalonia (Spain).

The criteria for subjects selection to participate in our project are:

1 . Inclusion criteria: patients with SLE according to established diagnostic criteria in 1997 2. Exclusion criteria:

* Presence of cardiac: Ischemic heart disease or congenital or acquired structural heart disease (hypertrophic cardiomyopathy, idiopathic dilated cardiomyopathy, valve disease with clinical significance).
* Background heart surgery or cardiac ablation procedures.
* Background in other pathological processes has been described affecting cardiac conduction tissue: Steinert's disease, Lyme disease, Chagas' disease with heart involvement or hypothyroidism.

The selection of patients and controls are done through a sampling of consecutive patients seen in our outpatient rheumatology center to achieve the sample size. This has been fixed in two subgroups: 100 patients with SLE and positive for anti-Ro (with positivity for anti-Ro only 52 or positivity for anti-Ro and anti-Ro 52 60) and 50 patients (controls ) with SLE and negative for anti-Ro (anti-Ro52 and anti-Ro 60).

As defined as primary variables, the study of cardiac conduction disorders will be done through the analysis of resting electrocardiogram (ECG) and a 24-hour Holter.

Other descriptive variables are listed below:

* Collection of general medical history of patients, with emphasis on Rheumatology and cardiac involvement.
* Check the current medication.
* Height and weight.
* Physical examination.
* 12-lead resting ECG with analysis of rate base, as well as the duration of the PR interval, QRS and QT. Analysis of the presence of intraventricular conduction disorders and the presence of ectopic beats.
* Record 24-hour Holter Presence and number of ventricular ectopic beats, classification of events according to the Lown's criteria. Presence of significant pauses (RR interval> 2000mseg). Measurement of corrected QT (QTc).
* Presence of autonomic dysfunction parameters: time domain parameters such as the mean RR interval, standard deviation of all normal RR intervals (SDNN), the root of the mean difference between successive adjacent normal RR intervals (RMSSD ) and the percentage of adjacent intervals over 50mseg (PNN50)
* Echocardiography to rule out structural heart disease: Analysis of ventricular diameters and systolic and diastolic function, presence of significant valve disease, pulmonary systolic pressure, pericardial effusion and other congenital or acquired structural heart disease.
* Analysis with serologic immune profile, determining the degree of organic involvement by SLE

ELIGIBILITY:
Inclusion Criteria:

* Patients with SLE diagnosis, according to SLE diagnostic criteria.

Exclusion Criteria:

* Patients with previous cardiac diseases (ischemic heart disease, hypertrophic cardiomyopathy, dilated cardiomyopathy, valvular heart disease)
* Clinical history of heart surgery or ablation procedures
* Clinical history of other conditions that affect heart conduction:

  * Steinert Disease
  * Lyme Disease
  * Chagas Disease
  * Hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SLE visited in the rheumatology outpatient's area.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Villuendas, Principal Investigator — GTIPUH
Locations (1):
- Germans Trias i Pujol University Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Background] Lazzerini PE, Capecchi PL, Laghi-Pasini F. Anti-Ro/SSA antibodies and cardiac arrhythmias in the adult: facts and hypotheses. Scand J Immunol. 2010 Sep;72(3):213-22. doi: 10.1111/j.1365-3083.2010.02428.x. PMID 20696018
- [Background] Chameides L, Truex RC, Vetter V, Rashkind WJ, Galioto FM Jr, Noonan JA. Association of maternal systemic lupus erythematosus with congenital complete heart block. N Engl J Med. 1977 Dec 1;297(22):1204-7. doi: 10.1056/NEJM197712012972203. PMID 917056
- [Background] Seferovic PM, Ristic AD, Maksimovic R, Simeunovic DS, Ristic GG, Radovanovic G, Seferovic D, Maisch B, Matucci-Cerinic M. Cardiac arrhythmias and conduction disturbances in autoimmune rheumatic diseases. Rheumatology (Oxford). 2006 Oct;45 Suppl 4:iv39-42. doi: 10.1093/rheumatology/kel315. PMID 16980722
- [Background] Edwards CS, Mootoo R, Bhanji A. High grade heart block in association with SLE. Ann Rheum Dis. 2004 May;63(5):606. doi: 10.1136/ard.2002.005322. No abstract available. PMID 15082501
- [Background] Costedoat-Chalumeau N, Georgin-Lavialle S, Amoura Z, Piette JC. Anti-SSA/Ro and anti-SSB/La antibody-mediated congenital heart block. Lupus. 2005;14(9):660-4. doi: 10.1191/0961203305lu2195oa. PMID 16218462
- [Background] Santos-Pardo I, Martinez-Morillo M, Villuendas R, Bayes-Genis A. Anti-Ro antibodies and reversible atrioventricular block. N Engl J Med. 2013 Jun 13;368(24):2335-7. doi: 10.1056/NEJMc1300484. No abstract available. PMID 23758256
- [Background] Behan WM, Behan PO, Gairns J. Cardiac damage in polymyositis associated with antibodies to tissue ribonucleoproteins. Br Heart J. 1987 Feb;57(2):176-80. doi: 10.1136/hrt.57.2.176. PMID 3493020
- [Background] Logar D, Kveder T, Rozman B, Dobovisek J. Possible association between anti-Ro antibodies and myocarditis or cardiac conduction defects in adults with systemic lupus erythematosus. Ann Rheum Dis. 1990 Aug;49(8):627-9. doi: 10.1136/ard.49.8.627. PMID 2396870
- [Background] O'Neill TW, Mahmoud A, Tooke A, Thomas RD, Maddison PJ. Is there a relationship between subclinical myocardial abnormalities, conduction defects and Ro/La antibodies in adults with systemic lupus erythematosus? Clin Exp Rheumatol. 1993 Jul-Aug;11(4):409-12. PMID 8403587
- [Background] Lodde BM, Sankar V, Kok MR, Leakan RA, Tak PP, Pillemer SR. Adult heart block is associated with disease activity in primary Sjogren's syndrome. Scand J Rheumatol. 2005 Sep-Oct;34(5):383-6. doi: 10.1080/03009740510026661. PMID 16234186
- [Background] Costa M, Gameiro Silva MB, Silva JA, Skare TL. Anti-RO anti-LA anti-RNP antibodies and eletrocardiogram's PR interval in adult patients with systemic lupus erythematosus. Acta Reumatol Port. 2008 Apr-Jun;33(2):173-6. PMID 18604183
- [Background] Lazzerini PE, Capecchi PL, Guideri F, Acampa M, Galeazzi M, Laghi Pasini F. Connective tissue diseases and cardiac rhythm disorders: an overview. Autoimmun Rev. 2006 May;5(5):306-13. doi: 10.1016/j.autrev.2005.11.002. Epub 2005 Dec 9. PMID 16782554
- [Background] Lazzerini PE, Capecchi PL, Acampa M, Morozzi G, Bellisai F, Bacarelli MR, Dragoni S, Fineschi I, Simpatico A, Galeazzi M, Laghi-Pasini F. Anti-Ro/SSA-associated corrected QT interval prolongation in adults: the role of antibody level and specificity. Arthritis Care Res (Hoboken). 2011 Oct;63(10):1463-70. doi: 10.1002/acr.20540. PMID 21739618
- [Background] Villuendas R, Olive A, Junca G, Salvador I, Martinez-Morillo M, Santos-Pardo I, Pereferrer D, Zamora E, Bayes-Genis A. Autoimmunity and atrioventricular block of unknown etiology in adults: the role of anti-Ro/SSA antibodies. J Am Coll Cardiol. 2014 Apr 8;63(13):1335-1336. doi: 10.1016/j.jacc.2013.10.086. Epub 2014 Jan 30. No abstract available. PMID 24486277
- [Background] Gordon PA, Rosenthal E, Khamashta MA, Hughes GR. Absence of conduction defects in the electrocardiograms [correction of echocardiograms] of mothers with children with congenital complete heart block. J Rheumatol. 2001 Feb;28(2):366-9. PMID 11246679
- [Derived] Villuendas R, Martinez-Morillo M, Junca G, Teniente-Serra A, Diez C, Heredia S, Riveros-Frutos A, Bayes-Genis A, Olive A. Usefulness of cardiac screening in patients with systemic lupus erythematosus and anti-Ro/SSA antibodies. Lupus. 2021 Sep;30(10):1596-1602. doi: 10.1177/09612033211027928. Epub 2021 Jul 1. PMID 34192953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SLE and Anti-Ro Antibodies Group | SLE Without Anti-Ro Antibodies Group
Started | 51 | 100
Completed | 46 | 99
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLE and Anti-Ro Antibodies Group | SLE Without Anti-Ro Antibodies Group | Total
Number analyzed (Participants) | 46 | 99 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.14 (11.75) | 45.24 (12.81) | 44.49 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 91 | 133
  Male | 4 | 8 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 42 | 91 | 133
  Ethnicity: Latin-American | 4 | 6 | 10
  Ethnicity: North-African | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Spain | 46 | 99 | 145

OUTCOME MEASURES:

1. Primary Outcome: Presence of Conduction Disorders in Patients With SLE Regarding to Its Serologic Profile
Description: Conduction disorders will be evaluated by 12-lead ECG recordings an 24-hour Holter recordings. Measurements will include PR intervals (in msec), QRS duration (in msec) .
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: msec
Groups:
- SLE and Anti-Ro Antibodies Group: Patients with SLE visited in the rheumatology outpatient's area with positivity to Anti-Ro antibodies. No intervention (only observational)
  No intervention: Observational
- SLE Without Anti-Ro Antibodies Group: Patients with SLE visited in the rheumatology outpatient's area with negativity to Anti-Ro antibodies. No intervention (only observational)
  No intervention: Observational
Arm/Group | SLE and Anti-Ro Antibodies Group | SLE Without Anti-Ro Antibodies Group
Number analyzed (Participants) | 46 | 99
msec
  QRS duration | 89.22 (8.5) | 91.41 (8.9)
  PR duration | 145.68 (21.1) | 146.72 (18.4)

2. Secondary Outcome: QT and Corrected QT Intervals
Description: Ventricular repolarization will be evaluated by 12-lead ECG recordings an 24-hour Holter recordings. Measurements will include QT and corrected QT intervals, and the presence of ventricular arrhythmia. Corrected QT (QTc) intervals will be obtained by measuring the QT interval (QTm) and the previous RR interval, following the Bazett formula (QTc=QTm divided by the square root of previous RR interval in seconds). A comparison will be made between the anti-Ro60 antibody positive patients and the anti-Ro60 antibody negative patients.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SLE and Anti-Ro Antibodies Group | SLE Without Anti-Ro Antibodies Group
Number analyzed (Participants) | 46 | 99
msec
  Corrected QT | 420.74 (24.3) | 421.33 (22.1)
  QT dispersion | 8.25 (7.8) | 6.81 (5.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | SLE and Anti-Ro Antibodies Group | SLE Without Anti-Ro Antibodies Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/99
Other Adverse Events (participants affected / at risk) | 0/46 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT02162992/Prot_SAP_ICF_000.pdf